CLINICAL TRIAL: NCT02622945
Title: Transcranial Direct Current Stimulation in Acute and Chronic Post-stroke Aphasia
Brief Title: Effects of Transcranial Direct Current Stimulation in Post-stroke Aphasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study could not recruit any participant
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NA00078932
Record Dates: First submitted 2015-11-17; First posted 2015-12-07 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS plus Speech-Language Therapy (Experimental): Active tDCS will be applied at the beginning of 45min speech-language therapy session and will last for 20 min. Language therapy will be oral and written naming. This is a cross-over study so all participants will receive this arm but the order will be randomized.
  Interventions: Device: Active tDCS plus Speech-Language Therapy
- Sham plus Speech-Language Therapy (Sham Comparator): Sham tDCS will be applied at the beginning of 45min speech-language therapy session. Language therapy will be oral and written naming. This is a cross-over study so all participants will receive this arm but the order will be randomized.
  Interventions: Device: Sham plus Speech-Language Therapy

INTERVENTIONS:
Device: Active tDCS plus Speech-Language Therapy — Stimulation will be delivered by a battery-driven constant current stimulator. The electrical current will be administered to a pre-specified region of the brain not affected by the lesion(perilesional areas, right hemisphere or cerebellum). The stimulation will be delivered at an intensity of 2mA (estimated current density 0.04 mA/cm2; estimated total charge 0.048C/cm2) in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will be oral and written naming.
  Other Names: Active tDCS and speech-therapy
  Arms: Active tDCS plus Speech-Language Therapy
Device: Sham plus Speech-Language Therapy — Speech-Language therapy will be administered during sham stimulation. Current will be administered in a ramp-line fashion but after the ramping the intensity will drop to 0 mA. Speech-language therapy will be oral and written naming.
  Other Names: Sham tDCS plus speech-therapy
  Arms: Sham plus Speech-Language Therapy

SUMMARY:
This study aims to determine whether transcranial direct current stimulation (tDCS) paired with speech-language therapy is more beneficial than speech-language therapy alone in acute and chronic post-stroke aphasia.

DETAILED DESCRIPTION:
This study aims to determine whether behavioral word-retrieval therapy coupled with anodal tDCS will improve the fluency and name retrieval performance of participants with post-stroke aphasia more efficiently and for greater duration than language therapy alone (i.e. in the sham condition).

tDCS neuronal targets will be selected in this order:

1. left posterior superior-middle temporal gyrus (an area critical for word retrieval and word comprehension),
2. left posterior frontal areas found to be responsible for lexical selection if the first area is infarcted, or
3. right cerebellum (important for learning, and consistently activated in naming task) if both of the other areas are infarcted.

The same areas will be stimulated during the first tDCS and sham periods. If the participant returns for a second period of tDCS and sham with language therapy, the right cerebellum will be stimulated (if it was the only uninfarcted target area investigators will stimulate this area again). For cerebellar stimulation, either anodal or cathodal will be used as studies show that anodal or cathodal stimulation has an effect on cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with with post-stroke aphasia and word-retrieval deficits
* Premorbid speakers of English
* Diagnosis will be based on neuropsychological testing, language testing (most commonly the Western Aphasia Battery), MRI and clinical assessment
* Stroke size: any l
* Location: Left hemisphere strokes only from any etiology.
* Time since stroke onset: 1 day to 20 years.

Exclusion Criteria:

* uncorrected visual or hearing impairment by self report
* other premorbid neurological disorder affecting the brain
* any other language-based learning disorder or other neurodegenerative disorder such as Alzheimer's Disease or Primary Progressive Aphasia
* premorbidly diagnosed with a developmental language disorder
* Pregnant women will also be excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in picture naming scores in trained and untrained items | Before and after 15 sessions of intervention (3 weeks) and at 2 weeks and 2 months follow-ups

SECONDARY OUTCOMES:
Change in Philadelphia Naming Test: Picture naming of everyday objects, different from training set | Before and after 15 sessions of intervention (3 weeks) and at 2 weeks and 2 months follow-ups
Change in Written naming of objects and actions | Before and after 15 sessions of intervention (3 weeks) and at 2 weeks and 2 months follow-ups
  The investigators will evaluate the absolute number as well as the percent change of the list of objects and actions assigned for intervention as trained and untrained items.
Change in working memory (digit span) | Before and after 15 sessions of intervention (3 weeks) and at 2 weeks and 2 months follow-ups
Change in verbal fluency | Before and after 15 sessions of intervention (3 weeks) and at 2 weeks and 2 months follow-ups
  The investigators will use letter (F, A, S) and semantic fluency measures (animals, fruits and vegetables) and the investigators will measure how many were added or omitted at follow-up intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Schlaug G, Marchina S, Wan CY. The use of non-invasive brain stimulation techniques to facilitate recovery from post-stroke aphasia. Neuropsychol Rev. 2011 Sep;21(3):288-301. doi: 10.1007/s11065-011-9181-y. Epub 2011 Aug 14. PMID 21842404
- [Background] Dmochowski JP, Datta A, Huang Y, Richardson JD, Bikson M, Fridriksson J, Parra LC. Targeted transcranial direct current stimulation for rehabilitation after stroke. Neuroimage. 2013 Jul 15;75:12-19. doi: 10.1016/j.neuroimage.2013.02.049. Epub 2013 Mar 5. PMID 23473936